CLINICAL TRIAL: NCT02059005
Title: Specialized Community Disease Management to Reduce Substance Use and Hospital Readmissions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCORI-1306-03482
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Drug Use; Alcohol Use; Congestive Heart Failure; Pneumonia; Acute Myocardial Infarction; Diabetes Mellitus; Chronic Obstructive Pulmonary Disease; End-Stage Renal Disease
Keywords: Addiction; Substance Use Disorder; Rehospitalization; Community Disease Management; Behavioral Health; Community Health Worker
MeSH Terms: conditions — Alcohol Drinking; Heart Failure; Pneumonia; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Kidney Failure, Chronic; Behavior, Addictive; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specialized Community Disease Management (Experimental): Specialized Community Disease Management
  Interventions: Behavioral: Specialized Community Disease Management
- Treatment As Usual (Active Comparator): Treatment as Usual: standard post-hospital discharge with medical monitoring.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Specialized Community Disease Management — Specialized Community Disease Management is 90-day program that employs specialized teams including a trained clinical social worker and a peer-specialist community health worker who provide evidence-based telephone continuing care, home visits, and focus on patients' substance use following hospital discharge.
  Arms: Specialized Community Disease Management
Behavioral: Treatment As Usual — Treatment as Usual is a 90-day, post-discharge program that consists of medical monitoring by nurses and community health workers who have no special training in working with substance use disorder patients, and does not address substance use.
  Arms: Treatment As Usual

SUMMARY:
This study will assess Specialized Community Disease Management (SCDM), an intervention which employs various evidence-based strategies to engage substance using co-morbid patients while in the hospital and follow them into the community via an empirically validated telephone approach as well as contact with a trained community health worker peer specialist. The investigators will first adapt and refine the core SCDM intervention with patient, provider, and stakeholder input through an active community advisory board. The investigators will then conduct a three-year, randomized controlled trial of 222 patients enrolled prior to hospital discharge who are diagnosed with congestive heart failure, pneumonia, acute myocardial infarction, chronic obstructive pulmonary disease, diabetes mellitus, or end-stage renal disease, and a substance use disorder (SUD). Patients will be randomized to either the SCDM intervention or Treatment as Usual (TAU), in which a team of nurse navigators and community health workers follow patients (primarily by telephone) for 90 days post-discharge, but do not address the specific needs of SUDs. The investigators will test the following four hypotheses: (1) patients randomized to SCDM will demonstrate larger reductions in substance use measured by urine-confirmed self-reported days using over the 6-month follow-up compared to patients randomized to TAU, (2) patients randomized to SCDM will attend more specialty substance abuse intervention and treatment sessions over the 6 month follow-up than patients randomized to TAU, (3) patients randomized to SCDM will demonstrate reduced HIV transmission risk behaviors and greater rates of HIV testing over the 6 month follow-up than patients randomized to TAU, and (4) patients randomized to SCDM will experience fewer days of rehospitalization and use of acute emergency services than patients randomized to TAU.

DETAILED DESCRIPTION:
Hospitalized patients with substance use disorders (SUDs) face significant complications in their medical care. They are more likely to be discharged against medical advice, rehospitalized after discharge, and experience personal chaos and reduced family support. Hospital systems are moving to implement hospital-based and community disease management strategies to help patients transition post-discharge, however, few provide specialized follow-up for patients with SUDs. This proposal will test whether an extended, specialized community disease management program can improve outcomes over an existing nurse navigator disease management strategy for patients with co-morbid medical conditions and SUDs. The investigators will enroll 222 inpatients with co-occurring medical conditions and SUDs and will randomly assign them to either 1) Treatment as Usual - a 90-day, post-discharge program that consists of medical monitoring by workers who have no special training in working with SUD patients, or 2) the Specialized Community Disease Management program - a 90-day program that will employ specialized teams including a trained clinical social worker and a peer-specialist community health worker who will provide evidence-based telephone continuing care, home visits, and increased focus on patients' substance use. All participants will be followed at 3- and 6-months post-discharge. The investigators hypothesize that (1) patients randomized to SCDM will demonstrate larger reductions in substance use measured by urine-confirmed self-reported days using over the 6-month follow-up compared to patients randomized to TAU, (2) patients randomized to SCDM will attend more specialty substance abuse intervention and treatment sessions over the 6 month follow-up than patients randomized to TAU, (3) patients randomized to SCDM will demonstrate reduced HIV transmission risk behaviors and greater rates of HIV testing over the 6 month follow-up than patients randomized to TAU, and (4) patients randomized to SCDM will experience fewer days of rehospitalization and use of acute emergency services than patients randomized to TAU.

ELIGIBILITY:
Inclusion Criteria:

* patient is 18 years or older
* alcohol and/or drug screening score that indicates at least mild problem severity

Exclusion Criteria:

* medical or psychiatric complications
* patient was admitted to hospital directly from a drug and alcohol inpatient rehabilitation facility
* patient reports plans to leave the area within the next 12 months
* patient is unable to provide valid informed consent
* patient is attending dialysis
* patient is not English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Brooks, PhD, Principal Investigator — Treatment Research Institute
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
in line with HIPAA protections, we will make our final dataset available to other researchers. Fully de-identified data will be available to any researcher. If a researcher should request a limited dataset then we will only share that data after obtaining an appropriate data use agreement which includes an agreement not to attempt to re-identify or contact participants. We will not share directly identifiable data with outside researchers per our HIPAA authorization for this study.

REFERENCES:
- See also: Patient-Centered Outcomes Research Institute Project Abstract — http://www.pcori.org/research-results/2013/specialized-community-disease-management-reduce-substance-use-and-hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Temple University Hospital between November 2015 and June 2016.
Pre-assignment Details: Participants were screened for eligibility using the AUDIT, DAST, and Mini-International Neuropsychiatric Interview (MINI) for substance use disorders.
Period: Overall Study
Arm/Group | Specialized Community Disease Management | Treatment As Usual
Started | 49 | 48
3 Month Assessment | 37 | 33
6 Month Assessment | 29 | 24
Completed | 29 | 24
Not Completed | 20 | 24
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 19 | 19
Not completed — Incarceration | 0 | 1
Not completed — Inpatient | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received a bedside SBIRT session following consent and randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Specialized Community Disease Management | Treatment As Usual | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.84 (7.71) | 48.65 (12.81) | 50.26 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 28 | 29 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 41 | 38 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 32 | 67
  White | 6 | 8 | 14
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97
Primary Substance of Use [Count of Participants; unit: Participants]
  Alcohol | 16 | 18 | 34
  Marijuana | 1 | 6 | 7
  Cocaine | 19 | 14 | 33
  Opioids | 5 | 2 | 7
  Other | 8 | 6 | 14
Index Medical Condition [Count of Participants; unit: Participants]
  Acute Myocardial Infarction | 1 | 4 | 5
  Congestive Heart Failure | 21 | 18 | 39
  Chronic Obstructive Pulmonary Disease | 6 | 8 | 14
  Diabetes | 5 | 4 | 9
  End Stage Renal Disease | 1 | 0 | 1
  Pneumonia | 4 | 1 | 5
  Rapid Rehospitalization | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Substance Use Rates From Baseline
Description: Urinalysis confirmed self-reported days of use for any substance, including alcohol, cocaine, marijuana, opiates, sedatives, and hallucinogens over time. Participants reported substance use for the 90 days prior to the assessment date.
Time Frame: 0, 3, 6 months
Population: The number analyzed in row differs from overall because the mixed-effects model analyses included participants who completed baseline and at least one follow-up. As a result, the number analyzed at each follow-up differed.
Measure: Mean (Standard Deviation); unit: Days of Substance Use
Arm/Group | Treatment As Usual | Specialized Community Disease Management
Number analyzed (Participants) | 48 | 49
Days of Substance Use
  Baseline | 51.37 (34.31) | 51.38 (31.77)
  3 Months: number analyzed (Participants) | 29 | 37
  3 Months | 35.53 (34.74) | 26.65 (32.9)
  6 Months: number analyzed (Participants) | 21 | 26
  6 Months | 30.65 (33.72) | 30.47 (36.30)

2. Secondary Outcome: Change in Treatment Session Attendance From Baseline
Description: Treatment sessions attended for alcohol or drug use issues over time. Participants self-reported attendance for the 6 months prior to the baseline assessment. During follow-up assessments, participants self-reported attendance since the last assessment date.
Time Frame: 0, 3, 6, months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days of attending treatment sessions
Arm/Group | Specialized Community Disease Management | Treatment As Usual
Number analyzed (Participants) | 45 | 48
Days of attending treatment sessions
  Baseline | 11.36 (24.78) | 4.75 (15.47)
  3 Months: number analyzed (Participants) | 35 | 27
  3 Months | 9.34 (22.75) | 5.93 (17.81)
  6 Months: number analyzed (Participants) | 23 | 22
  6 Months | 6.17 (19.48) | 3.27 (7.03)

3. Secondary Outcome: Number of Hospitalizations and Use of Emergency Services
Description: Days of hospitalization and days of use of acute emergency services after Baseline. Participants self-reported their service utilization for the 6 months prior to the baseline assessment. During follow-up assessments, participants self-reported their service utilization since the last assessment date.
Time Frame: 0, 3, 6, months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days of ER or Hospital Utilization
Arm/Group | Specialized Community Disease Management | Treatment As Usual
Number analyzed (Participants) | 45 | 42
Days of ER or Hospital Utilization
  Baseline | 3.53 (4.79) | 5.5 (10.55)
  3 Months: number analyzed (Participants) | 33 | 23
  3 Months | 4.76 (8.81) | 4.91 (10.91)
  6 Months: number analyzed (Participants) | 23 | 22
  6 Months | 4.17 (4.86) | 3.55 (9.83)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious Adverse Events were defined as death; a life threatening event such as suicidal ideation/attempt or inpatient rehospitalization related to the index medical condition, suicidal behavior, psychiatric distress, or drug/alcohol complications/overdose. Unrelated medical events that did not require hospitalization were not be considered SAEs.
Arm/Group | Specialized Community Disease Management | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 1/49 | 3/48
Serious Adverse Events (participants affected / at risk) | 23/49 | 14/48
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Specialized Community Disease Management (N=49) | Treatment As Usual (N=48)
Hospitalization for congestive heart failure (Cardiac disorders) | 9 (23) | 7 (15)
Hospitalization for COPD (Respiratory, thoracic and mediastinal disorders) | 6 (13) | 4 (5)
Hospitalization for Diabetes (Renal and urinary disorders) | 2 (5) | 2 (4)
Hospitalization for end-stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hospitalization for pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hospitalization for cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Suicidal ideation/attempt (Psychiatric disorders) | 2 (2) | 3 (3)
Hospitalization for Syncope (General disorders) | 1 (1) | 0 (0)
Hospitalization for drug/alcohol use (Psychiatric disorders) | 1 (1) | 0 (0)
Inpatient Drug/Alcohol (Psychiatric disorders) | 1 (1) | 1 (1)
Death, Cause Unknown (General disorders) | 1 (1) | 1 (1)
Death related to congestive heart failure (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT02059005/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT02059005/SAP_001.pdf
  • Informed Consent Form (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT02059005/ICF_002.pdf